CLINICAL TRIAL: NCT04129229
Title: Non-Randomized, Multi-Site, Single-Arm Study of the LinguaFlex™ Tongue Retractor (LTR) for the Treatment of Moderate to Severe Obstructive Sleep Apnea and Snoring in Adult Subjects
Brief Title: LinguaFlex Tongue Retractor (LTR) for the Treatment of OSA and Snoring in Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Linguaflex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTR-006-V02.0-US-CTP
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea; Snoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- LTR Treatment (Experimental): Eligible subjects will undergo insertion of the LTR device in their tongue. Initiation of treatment will occur 7 days post insertion procedure and will be monitored over the course of 1 year.
  Interventions: Device: LinguaFlex Tongue Retractor (LTR)

INTERVENTIONS:
Device: LinguaFlex Tongue Retractor (LTR) — The LinguaFlex Tongue Retractor (LTR) is a small, flexible, implanted tongue retaining device that lessens the backward movement of the tongue during sleep. The LTR's flexible shaft and a nubbed tether passes through the center of the tongue beneath the tongue blade (frenulum area) and connects to a disc (head) that rests on the external surface of the tongue base mucosa. Underneath the tongue, on the external surface of the frenulum, a small anchor secures the shaft that can be adjusted to tension the LTR to maximize therapeutic effect and maintain comfort.

SUMMARY:
The LinguaFlex™ Tongue Retractor (LTR) is an investigational medical device that is inserted into the tongue to lessen its backward movement during sleep. This helps to keep the airway open during sleep so that the tongue doesn't block the airway causing obstructive apnea or narrow it enough to cause snoring. This study will monitor the effectiveness of the LTR device in the reduction of Obstructive Sleep Apnea and snoring over the course of a one-year treatment period.

DETAILED DESCRIPTION:
The study design is a multi-site, prospective, open-label, non-randomized, single-arm clinical study to test the efficacy of the LinguaFlex Tongue Retractor for the treatment of moderate to severe Obstructive Sleep Apnea (OSA) (AHI ≥15 at baseline) in adult subjects in twelve (12) months of continuous use. The study will include three (3) investigational sites that will implant a maximum of eighty (80) subjects with the LTR. No single site is to perform more than 35 implants. After informed consent is obtained, eligible subjects (adults who have moderate to severe OSA) will be screened for study inclusion. The screening will consist of a Home Sleep Test (HST) completed within four (4) months of inclusion in the study to confirm the diagnosis of moderate to severe OSA, an Epworth Sleepiness Scale (ESS) assessment, Snoring Self-Assessment (SOS) with bed partner input (SBPS), assessment of pain, speech and swallowing, and a physical examination. The screening data will be reviewed by the Sponsor's designated study monitor to confirm and approve that inclusion criteria are fully met. Failure to meet all inclusion criteria will be designated as a screen failure and the subject's enrollment will be terminated. Participation in the study is voluntary. Subjects may withdraw at any time during the study. Reasons for the withdrawal will be recorded and entered into the clinical study report. Any subject who withdraws from the study for any reason will have the device removed and will undergo a Post Device Removal Follow-Up within 30 days (-7/+ 15) of device removal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects able to read, understand and sign consent
* Subjects 18 years or older with:

  1. Moderate to severe OSA (AHI of ≥ 15 to ≤ 50 as determined by a Diagnostic PSG recording within 2 months of inclusion)
  2. Subject agrees not to use any type of additional OSA therapy including PAP therapy throughout the course of the study

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation in the clinical trial:

* < 18 years of age
* AHI < 15(mild OSA)
* AHI > 50
* Subjects with > 20% of AHI score accounted for from central apnea
* More than 10% of Total Sleep Time (TST) with blood O2 saturation (SaO2) below 70%
* Subjects successfully treated with prescribed PAP therapy
* Tonsillar hypertrophy ≥3
* Subjects with significant active comorbid respiratory or cardiac disease (such as COPD or Heart Failure)
* Subjects requiring regular use of supplemental oxygen
* Nasal airway obstruction as seen on examination
* Congenital malformations of the upper airway, larynx, pharynx, oral cavity or tongue
* Narrowing of hypopharynx airspace more than velopharyngeal airspace as seen on examination (suspected epiglottic obstruction)
* History of radiation therapy to the neck or upper respiratory tract
* Subjects with bleeding disorders, unresolved impaired immunity for any reason, or heart attack within the last six months
* Subjects with an existing tongue stud/piercing
* Females who are pregnant (anesthesia risk)
* Allergy to LTR materials (Silicone, PEEK, Polyurethane)
* Subjects who have in the surgeon's judgment unusual anatomy that would interfere with treatment or increase the risk for the procedure
* Unable and/or unwilling to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Responder to Therapy | One Year
  Determine the responder rate to therapy. A responder is defined as a subject who experiences a ≥ 50% reduction in AHI from baseline and has an AHI < 20 at the 12-month follow-up visit. Subjects with an AHI ≤ 20 at baseline will be considered a responder if a 50% reduction in AHI is achieved from baseline.

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale (ESS) | One Year
  Determine the change in Epworth Sleepiness Scale (ESS) from the baseline control measurement and determine the proportion of study subjects that achieve an ESS value of ≤ 10 at the twelve-month follow-up. ((ESS is a validated instrument that rates a subject's daytime sleepiness and is commonly used in clinical evaluation and management of OSA as a quality of life measurement. Scores range from 0 to 24, with lower scores indicating greater functioning. An ESS < 10 is considered normal subjective sleepiness.)
Oxygen Desaturation Index (ODI) Responder | One Year
  Determine the Oxygen Desaturation Index (ODI) responder rate at the twelve-month follow-up visit. An ODI responder is defined as a subject which demonstrates at least a 25% reduction in ODI from the baseline control measurement at the 12-month follow-up visit. Change in ODI will be reported as a percentage change from baseline for each subject as well as the mean percentage change for the entire cohort.

OTHER OUTCOMES:
Quality of Life Metric - Pain | At each follow-up visit over the course of 1 year
  Examine the tolerance and comfort of the implanted LTR. Pain will be assessed at each follow-up visit using a 10 point Visual Analog Scale (0 no pain - 10 worst pain) and will be compared to the baseline measurement.
Quality of Life Metric - Speech and Swallowing | At each follow-up visit over the course of 1 year.
  Examine the tolerance and comfort of the implanted LTR. Comfort with speech and swallowing will be assessed using the Performance Status Scale for Head and Neck Cancer Patients (PSS-HN). This scale consists of three individual scores for Normalcy of Diet, Eating in Public and Understanding of Speech. In each case a score of 100 indicates normal function and 0 indicates the most limited function.
Quality of Life Metric - Snoring | At each follow-up visit over the course of 1 year.
  Examine the change in snoring from the baseline control measurement. Snoring will be assessed using the Snore Outcome Survey (SOS) and the Spouse/Bed Partner Survey (SBPS). The SOS is a series of 8 questions with a score range of 0 - 100; with 0 representing the worst possible snoring and 100 representing no snoring. The Spouse Bed Partner Survey is a series of 3 questions with a score range of 0 - 100; with a score of 0 representing the worst possible snoring and 100 representing no snoring.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Sanders, MD, Study Director — Linguaflex, Inc.
Locations (3):
- United States (3):
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - WVU Medicine / J. W. Ruby Memorial Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.